CLINICAL TRIAL: NCT05281627
Title: Psycho-Social Outcomes Following Emergency Laparotomy
Acronym: POLO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: NHS Greater Glasgow and Clyde (Other); The Royal College of Surgeons of England (Other)
Responsible Party: Sponsor
Other Study IDs: 8160
Record Dates: First submitted 2021-11-29; First posted 2022-03-16 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-03

CONDITIONS: Emergency Laparotomy
Keywords: Emergency Laparotomy; Laparotomy; Surgical Outcomes; Psychosocial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Emergency Laparotomy Patients: All adult patients (18+) who have undergone Emergency Laparotomy surgery, are recovering well (no illness which is expected to limit life to <6m post op) and have sufficient English-language and cognitive skills to complete the study questionnaires.
  Interventions: Other: Emergency Laparotomy
- Family Caregivers: Adult (18+) family members, close friend or caregivers of the individual who has received EmLap treatment have sufficient English-language and cognitive skills to complete the study questionnaires.

INTERVENTIONS:
Other: Emergency Laparotomy — All patients undergoing Emergency Laparotomy
  Groups: Emergency Laparotomy Patients

SUMMARY:
An emergency laparotomy (EmLap) is a life-saving operation; but the aftermath for those that do survive can be lifechanging. Each year, in excess of 25,000 EmLaps are performed in UK. A national effort, through the National Emergency Laparotomy Audit (NELA), has managed to improve peri-operative care, and reduce 30 day mortality from 1 in 4 to less than 1 in 10. Whilst this reduction should be commended, it also means that more patients are surviving with some form of new infirmity.

This infirmity may be short-lived and reversible in some, and yet others may transition into a permanent chronic disease state. The impact of EmLap on those individuals that "do not fully recover" is far-reaching and often interlinked, covering biological, social and psychological domains. This makes it difficult to describe the true problem, i.e. holistic morbidity and suggest an intervention to improve it.

The primary aim of this work is to describe the holistic morbidity of EmLap throughout the first year of a patient's recovery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above
* Able to communicate in English
* Cognitively able to complete the questionnaire
* Able to provide informed voluntary consent
* Undergone an EmLap during admission
* Clinical team anticipate to be "medically fit for discharge" within 48 hours (of consent)

Exclusion Criteria:

* Any terminal diagnosis in which the clinical team do not anticipate life expectancy to exceed 6 months from the time of surgery
* Acutely unwell at the time of recruitment. These patients may still be eligible and can be re-screened and recruited at a later date, should their condition improve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is all patients who have undergone emergency laparotomy during their admission to hospital, are recovering well and approaching discharge. Participants will be recruited from hospital sites in Wales and Scotland.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The change in patient reported Quality of Life as assessed by the EuroQuol 5-Dimension Health-related Quality of Life instrument (EQ-5D) | 12 months
  Patient reported Quality of Life will be measured at 3 time points post-discharge. Reduction of EQ-5D 3-Level scale (min.5; max 15) and EQ-5D Visual Analogue Scale (min 0; max. 100) represent improved quality of life.

SECONDARY OUTCOMES:
Establishing the patient definition of 'Recovery' following Emergency Laparotomy using qualitative methods | 12 months
  Semi-structured qualitative interviews will be conducted with approximately 15 Emergency Laparotomy patients, at 6-months post-discharge from hospital. The interview will evaluate:
  A) what patients consider to constitute 'recovery' following emergency laparotomy B) what factors influence achieving 'recovery' C) the timelines linked to a) and b)
Change in Fatigue Severity Score | 12 months
  Fatigue severity score (FSS) to assess physical health. Measured at 3 time-points post-operatively and scored from 9 (min.) to 63 (max.), with increase in total score represents greater fatigue severity/ reduced physical health.
Change in Body Mass Index | 12 months
  Body Mass Index (BMI) to assess physical health. Weight and Height will be recorded in kg and cm (respectively) at 3 time-points and BMI will be calculated and reported in terms of kg/m^2.
Change in Rockwood Frailty Score | 12 months
  Rockwood Frailty Score to asses physical health. Collected at 3 time-points and scored from 1 (min.) to 9 (max.), where greater score represents increased frailty. Only validated for use in the over 65's
Change in Gastro-Intestinal Quality of Life Index | 12 months
  Gastro-intestinal Quality of Life Index (GIQLI) to assess in physical health. Collected at 3 time-points, total score calculated from 0 (min.) to 144 ( max.), where greater total score represents improved GI health related QoL.
Change in International Trauma Questionnaire score | 12 months
  International Trauma Questionnaire to assess mental-health. Collected at 3 timepoints. Scored in accordance with assessment guidance to determine clinical signs of (complex) Post-Traumatic Stress Disorder.
Change in Patient Health Questionnaire score | 12 months
  Patient Health Questionnaire (PHQ9) to assess mental-health. Collected at 3 timepoints and scored from 0 (min.) to 27 (max.), where greater score represents increased depression severity.
Change in Generalised Anxiety Disorder assessment score | 12 months
  Generalised Anxiety Disorder assessment (GAD7) to assess mental-health. Measured at 3 timepoints from 0 (min.) to 21 (max.), where greater score represents increased anxiety severity.
Changes in Community Integration Questionnaire score | 12 months
  Community Integration Questionnaire (CIQ) to determine changes in social integration. Scored between 0 (min.) and 35 (max.), where greater score represents reduced social integration.
Change in sexual function | 12 months
  Single question regarding change in sexual function (min 0; max 5), where greater score represents increased sexual impairment
Change in employment status | 12 months
  Single question regarding change in employment status (yes/no).
The changes in care burden as assessed by the Modified Caregiver Strain Index (MCSI) | 12 months
  Caregiver- reported burden will be measured at 3 timepoints post-discharge. Increase in total score of the Modified Caregiver Strain Index (MCSI) (min. 0; max. 26), represents greater burden on caregiver.

OTHER OUTCOMES:
Overall patient experience of Emergency Laparotomy care as assessed by the NHS Wales Experience Questionnaire | 12 months
  Patient experience will be assessed at a 3 time-points during the course of their recovery at the end of the study using the NHS Wales Patient Experience questionnaire. Overall experience is measured on 10-point Likert scale (0-least satisfied, 10 most satisfied).
Number of patient points of care | 12 months
  Incidence of scheduled and unscheduled care will be measured over the course of the patients involvement in the project

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Alexandra Hospital, Paisley, Renfrewshire
  - Julie Cornish, Cardiff

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva L, Abbas Mohamed S, Meggy A, Ng JH, Torkington J, Moug S, Watts T, Bisson J, Cornish JA. Psychosocial outcomes following emergency laparotomy (POLO) study: a study protocol for a multicentre mixed-methods prospective cohort study assessing the psycho-social outcomes following emergency laparotomy in adults. BMJ Open. 2024 Jul 9;14(7):e081821. doi: 10.1136/bmjopen-2023-081821. PMID 38986553